CLINICAL TRIAL: NCT02314442
Title: A Phase 1, Randomized, Single Blind, Placebo Controlled, Single Ascending Dose and Multiple Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Subcutaneously Administered ALN PCSSC in Subjects With Elevated Low Density Lipoprotein Cholesterol
Brief Title: A Phase 1 Study of an Investigational Drug, ALN-PCSSC, in Subjects With Elevated Low Density Lipoprotein Cholesterol (LDL-C)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alnylam Pharmaceuticals (Industry)
Collaborators: The Medicines Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ALN-PCSSC-001
Record Dates: First submitted 2014-12-05; First posted 2014-12-11 (Estimated); Last update posted 2015-12-17 (Estimated); Status verified 2015-12

CONDITIONS: Hypercholesterolemia
Keywords: LDL-C; RNAi therapeutic
MeSH Terms: conditions — Hypercholesterolemia | interventions — ALN-PCS

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- ALN-PCSSC (Active Comparator)
  Interventions: Drug: ALN-PCSSC
- Sterile Normal Saline (0.9% NaCl) (Placebo Comparator)
  Interventions: Drug: Sterile Normal Saline (0.9% NaCl)

INTERVENTIONS:
Drug: ALN-PCSSC — Single or multiple doses of ALN-PCSSC by subcutaneous (sc) injection
  Arms: ALN-PCSSC
Drug: Sterile Normal Saline (0.9% NaCl) — calculated volume to match active comparator
  Arms: Sterile Normal Saline (0.9% NaCl)

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of ALN-PCSSC in subjects with elevated LDL-C.

ELIGIBILITY:
Inclusion Criteria:

* Adequate complete blood counts, liver and renal function
* Female subjects must be of non-childbearing potential; e.g. post-menopausal or pre-menopausal with surgical sterilization
* Male subjects agree to use appropriate contraception
* Willing to provide written informed consent and willing to comply with study requirements.
* Non-smokers and non-nicotine users for at least 90 days before screening
* On stable statin co-medication [for designated multiple dose cohorts only]

Exclusion Criteria:

* Any uncontrolled or serious disease, or any medical or surgical condition, that may interfere with participation in the clinical study and/or put the subject at significant risk
* Received an investigational agent within 90 days before the first dose of study drug or are in follow-up of another clinical study
* History of multiple drug allergies or intolerance to subcutaneous injection
* Received any medication or nutraceutical to alter serum lipids within 30 days before screening (non-statin cohorts only)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2014-12; Primary Completion 2015-05 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
The safety of ALN-PCSSC evaluated by the proportion of subjects experiencing adverse events (AEs), serious adverse events (SAEs), and AEs leading to study drug discontinuation | Part 1 (SAD phase): up to 180 days post dose; Part 2 (MD) phase: up to 180 days post final dose

SECONDARY OUTCOMES:
The pharmacokinetics (PK) of ALN-PCSSC (Cmax, tmax, AUC, t1/2) | Part 1 (SAD) phase: predose, 0.5,1,2,4,6,8,12,24,48,72,96 hours; 7, 14, 21, 28, 42, 56 days post-dose; Part 2 (MD) phase: predose, 0.5,1,2,4,6,8,12,24,48,72,96 hours; 7, 14, 21, 28, 29, 35, 42, 56, 84 days post-dose
The effect of ALN-PCSSC on serum levels of LDL-C | Through the sooner of final follow up visit or 180 days post final dose
The effect of ALN-PCSSC on plasma levels of PCSK9 | Through the sooner of final follow up visit or 180 days post final dose

CONTACTS AND LOCATIONS:
Overall Officials: Robert Kauffman, MD, Study Director — Alnylam Pharmaceuticals
Locations (2):
- United Kingdom (2):
  - Covance Clinical Research Unit, Leeds
  - Richmond Pharmacology, London

REFERENCES:
- [Derived] Fitzgerald K, White S, Borodovsky A, Bettencourt BR, Strahs A, Clausen V, Wijngaard P, Horton JD, Taubel J, Brooks A, Fernando C, Kauffman RS, Kallend D, Vaishnaw A, Simon A. A Highly Durable RNAi Therapeutic Inhibitor of PCSK9. N Engl J Med. 2017 Jan 5;376(1):41-51. doi: 10.1056/NEJMoa1609243. Epub 2016 Nov 13. PMID 27959715